CLINICAL TRIAL: NCT01107561
Title: Incision-first Versus Classic Seldinger Technique for Emergency Cricothyroidotomy
Brief Title: Different Techniques for Emergency Cricothyroidotomy
Acronym: CRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Association of Emergency Physicians (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00011192
Record Dates: First submitted 2010-04-12; First posted 2010-04-21 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Intubation, Intratracheal
Keywords: cricothyroidotomy; intubation; airway; emergency medicine; education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Seldinger technique (Experimental): Involves blind needle insertion through the skin into the cricoid membrane followed by insertion of the guide-wire and subsequent insertion of the tube over the guidewire.
  Interventions: Other: Seldinger technique
- Surgical airway approach (Active Comparator): The classical open or surgical technique involves a vertical skin incision with blunt dissection and identification of the anatomy followed by incision of the cricoid membrane and tube insertion.
  Interventions: Device: Surgical Airway Approach

INTERVENTIONS:
Other: Seldinger technique — Involves blind needle insertion through the skin into the cricoid membrane followed by insertion of the guide-wire and subsequent insertion of the tube over the guidewire
  Other Names: Neddle approach
  Arms: Seldinger technique
Device: Surgical Airway Approach — The classical open or surgical technique involves a vertical skin incision with blunt dissection and identification of the anatomy followed by incision of the cricoid membrane and tube insertion.
  Other Names: Open approach
  Arms: Surgical airway approach

SUMMARY:
This educational study will examine two different techniques for training emergency residents and staff on achieving a surgical airway (called a cricothyroidotomy).

DETAILED DESCRIPTION:
Introduction: In patients that cannot be intubated or ventilated by conventional means an emergency cricothyroidotomy is a potentially life saving intervention that is the common final pathway of difficult airway algorithms. Significant debate surrounds the ideal method of performing an emergency cricothyroidotomy. The literature remains divided between the open (surgical) and closed (wire assisted, or Seldinger) techniques. We feel that these two methods are not mutually exclusive and are proposing a novel "incision first" modification to the traditional Seldinger closed technique. Making a small (1 cm) incision prior needle insertion could facilitate localization of landmarks and may improve speed or success rate of the closed Seldinger procedure.

Introduction: In patients that cannot be intubated or ventilated by conventional means an emergency cricothyroidotomy is a potentially life saving intervention that is the common final pathway of difficult airway algorithms. Significant debate surrounds the ideal method of performing an emergency cricothyroidotomy. The literature remains divided between the open (surgical) and closed (wire assisted, or Seldinger) techniques. We feel that these two methods are not mutually exclusive and are proposing a novel "incision first" modification to the traditional Seldinger closed technique. Making a small (1 cm) incision prior needle insertion could facilitate localization of landmarks and may improve speed or success rate of the closed Seldinger procedure.

Methods: Using concealed allocation, this randomized controlled cross-over trial will be performed in a laboratory setting. Outcome assessment will be blinded. Both staff and resident emergency physicians will be included in this trial. We will use a well-validated swine trachea model for this study.

Results: Results will be collected using standardized Case Report Forms (CRF) and independently entered into a pre-constructed Microsoft ACCESS database. The primary outcome will be time to procedure completion. Secondary outcomes will be proportion of successful cricothyroidotomy, complications and ease of procedure and ability to increase clinical confidence using this model. Paired t-tests and Fisher's exact test will be used to compare the outcomes and due to multiple statistical tests, a correction will be used to adjust for multiple tests (p < 0.025) to indicate significance.

Conclusions: This study will assess and evaluate both the incision first model and closed Seldinger cricothyroidotomy techniques. We will discuss the merits of each technique and the effectiveness of the model.

ELIGIBILITY:
Inclusion Criteria:

All staff and residents presenting to a airway lab for Informed verbal consent.

Exclusion Criteria:

Non-physicians

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Time to complete airway access | Within the 5 minutes permitted for each procedure
  Measured in seconds as the time taken for insertion of the tube and connection of the bagging device.

SECONDARY OUTCOMES:
Success | Within 5 minutes of the start of the procedure
  Will be confirmed by inspection of the catheter within the tracheal lumen post procedure.
Number of attempts | Within the 5 minutes permitted for each procedure
  Number of needle insertions, sweeps with blade, guide-wire insertions, dilatation attempts and catheter insertions attempts.
Complications | Within the 5 minutes permitted for each procedure
  Penetration of posterior wall or placement of the tube outside the trachea
Perceived difficulty | Prior to end of the educational session
  Self-completed survey/questionnaire to assess level of difficulty and preference.

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Dong, MD, MSc, Principal Investigator — University of Alberta; Warren Thirsk, MD, FRCPC, Principal Investigator — University of Alberta; Brian H Rowe, MD, MSc, Study Director — University of Alberta; Cristina Villa-Roel, MD, MSc, Study Director — University of Alberta
Locations (1):
- Department of Emergency Medicine, Edmonton, Alberta, Canada